CLINICAL TRIAL: NCT02243553
Title: Evaluating the Effects of Tipranavir (With Ritonavir) Capsule and Liquid Formulation on Cytochrome P450 and P-glycoprotein Activity Using a Biomarker Cocktail in Healthy Human Volunteers
Brief Title: Effects of Tipranavir (With Ritonavir) Capsule and Liquid Formulation on Cytochrome P450 and P-glycoprotein Activity in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.101
Record Dates: First submitted 2014-09-01; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Caffeine; Warfarin; Vitamin K; Omeprazole; Dextromethorphan; Midazolam; Digoxin

ARMS (4):
- Treatment A (Experimental): tipranavir (TPV) capsule + ritonavir (RTV) capsule + cocktail + digoxin oral
  Interventions: Drug: Tipranavir capsule; Drug: Ritonavir capsule; Drug: Caffeine; Drug: Warfarin sodium; Drug: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Midazolam injection; Drug: Midazolam oral solution; Drug: Digoxin tablet
- Treatment B (Experimental): TPV capsule + RTV capsule + cocktail + digoxin injection
  Interventions: Drug: Tipranavir capsule; Drug: Ritonavir capsule; Drug: Caffeine; Drug: Warfarin sodium; Drug: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Midazolam injection; Drug: Midazolam oral solution; Drug: Digoxin injection
- Treatment C (Experimental): TPV solution + RTV capsule + cocktail + digoxin oral
  Interventions: Drug: Tipranavir solution; Drug: Ritonavir capsule; Drug: Caffeine; Drug: Warfarin sodium; Drug: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Midazolam injection; Drug: Midazolam oral solution; Drug: Digoxin tablet
- Treatment D (Experimental): TPV solution + RTV capsule + cocktail + digoxin injection
  Interventions: Drug: Tipranavir solution; Drug: Ritonavir capsule; Drug: Caffeine; Drug: Warfarin sodium; Drug: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Midazolam injection; Drug: Midazolam oral solution; Drug: Digoxin injection

INTERVENTIONS:
Drug: Tipranavir capsule
  Arms: Treatment A; Treatment B
Drug: Tipranavir solution
  Arms: Treatment C; Treatment D
Drug: Ritonavir capsule
Drug: Caffeine
Drug: Warfarin sodium
Drug: Vitamin K
Drug: Omeprazole
Drug: Dextromethorphan hydrobromide
Drug: Midazolam injection
Drug: Midazolam oral solution
Drug: Digoxin tablet
  Arms: Treatment A; Treatment C
Drug: Digoxin injection
  Arms: Treatment B; Treatment D

SUMMARY:
Primary: To quantify the influence of single-dose and steady-state tipranavir/ritonavir 500/200 mg on intestinal and hepatic cytochrome P450 (CYP) and P-glycoprotein (P-gp) biomarkers, as a means of predicting drug interactions. The AUCs for biomarkers caffeine, warfarin, omeprazole, dextromethorphan, midazolam, and digoxin will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Healthy subjects aged between 18 years and 45 years inclusive
3. Weighing at least 50 kg
4. Volunteers must be hospitalized on Days 1-4, 7-9, and 17-20 for pharmacokinetic assessments for each biomarker and TPV/r (Days 7-9 and 17-20)
5. Volunteers must be willing to complete all study-related activities
6. Each volunteer must have a valid social security number
7. Each volunteer must have acceptable medical history, physical examination and laboratory test

Exclusion Criteria:

1. History or presence of allergy to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
2. Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
3. History or diagnosis of any significant medical conditions: Including but not limited to gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hematological, psychiatric, neurological, oncological or hormonal disorders
4. Known elevated liver enzymes in past clinical trials with any compound (experimental or marketed)
5. Clinically relevant laboratory abnormalities (e.g. Hgb<11g/dL, Hct<30g/dL, total cholesterol >240mg/dL, triglycerides >500mg/dL, fasting glucose >130mg/dL, liver function tests >2.5x upper limit of normal, baseline international normalized ratio >1.2)
6. History of evidence of clinically significant hepatic, cardiac, pulmonary, endocrine, immunological, gastrointestinal, hematological, vascular or collagen disease
7. History of alcohol abuse or use of any illicit drugs
8. Unable to abstain from more than one beer or alcohol equivalent per day for the duration of the study
9. Use of tobacco products and/or history of smoking within the past 2 months
10. Pregnant or breast feeding
11. Sexually active women of childbearing age who do not use an acceptable barrier method of birth control
12. Hypersensitivity to caffeine, warfarin, vitamin K, omeprazole, dextromethorphan, midazolam, tipranavir, ritonavir or their excipients
13. Concomitant treatment with other experimental compounds
14. Concomitant administration of any prescription or over the counter medications known to alter P450 enzyme or P-gp activity
15. Concomitant administration of any prescription or over the counter medications known to be highly dependent on P450 or P-gp for clearance for which elevated plasma concentrations are known to be associated with serious toxicity
16. Concomitant administration of any food product known to alter P450 enzyme or P-gp activity such as grapefruit juice, Seville oranges
17. Concomitant administration of any drug that could affect bleeding (e.g., aspirin, clopidogrel, ticlopidine, warfarin, heparin, low-molecular weight heparin)
18. Concomitant administration of oral contraceptives (may be included with 7-day washout period)
19. Concomitant administration of any herbal medications
20. Inadequate venous access
21. Renal or hepatic insufficiency
22. Clinically unacceptable result at the screening physical examination
23. Use of investigational medications within 30 days before study entry
24. HIV-positive
25. Body Mass Index (BMI) > 30 kg/m²

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-01; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC) at steady state | up to 72 hours

SECONDARY OUTCOMES:
Plasma concentration after 12 hours (Cp12h) | 12 hours
Maximum plasma concentration (Cmax) | up to 12 hours
Time of maximum concentration (Tmax) | up to 72 hours
Apparent terminal half-life (t1/2) | up to 72 hours
Area under plasma concentration-time curve (AUC) after single dose | up to 72 hours
Change in biomarkers | baseline, up to 22 days
Change in enzyme activity | baseline, up to 22 days